CLINICAL TRIAL: NCT00265018
Title: HD10 for Early Stages
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HD10
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Hodgkin´s Lymphoma
Keywords: Hodgkin´s lymphoma; early stages
MeSH Terms: interventions — Doxorubicin; Bleomycin; Vinblastine; Dacarbazine

ARMS (4):
- Arm A (Active Comparator)
  Interventions: Drug: Adriamycin; Drug: Bleomycin; Drug: Vinblastine; Drug: DTIC; Radiation: 30 Gy IF-RT
- Arm B (Experimental)
  Interventions: Drug: Adriamycin; Drug: Bleomycin; Drug: Vinblastine; Drug: DTIC; Radiation: 20 Gy IF-RT
- Arm C (Experimental)
  Interventions: Drug: Adriamycin; Drug: Bleomycin; Drug: Vinblastine; Drug: DTIC; Radiation: 30 Gy IF-RT
- Arm D (Experimental)
  Interventions: Drug: Adriamycin; Drug: Bleomycin; Drug: Vinblastine; Drug: DTIC; Radiation: 20 Gy IF-RT

INTERVENTIONS:
Drug: Adriamycin
Drug: Bleomycin
Drug: Vinblastine
Drug: DTIC
Radiation: 30 Gy IF-RT
  Arms: Arm A; Arm C
Radiation: 20 Gy IF-RT
  Arms: Arm B; Arm D

SUMMARY:
This study is designed to find the optimum radiation dose and number of cycles for an ABVD chemotherapy combined with an involved field irradiation. It is to be tested whether the reduction from 4 to 2 cycles of ABVD and/or the reduction of the radiation dose from 30 to 20 Gy is feasible without a loss of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin´s lymphoma (histologically proven)
* CS (PS) IA, IB, IIA,IIB without any of the following risk factors:

  1. bulky mediastinal mass (> 1/3 maximum transverse thorax diameter)
  2. extranodal involvement
  3. ESR > 50 (A), > 30 (B-symptoms)
  4. 3 or more lymph node areas involved
* written informaed consent

Exclusion Criteria:

* Leukocytes <3000/microl
* Platelets <100000/microl
* Hodgkin´s Disease as "composite lymphoma"
* Activity index (WHO) < grade 2

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1370 (Actual)
Dates: Start 1998-05; Primary Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Volker Diehl, Prof., Principal Investigator — University of Cologne

REFERENCES:
- [Result] Engert A, Plutschow A, Eich HT, Lohri A, Dorken B, Borchmann P, Berger B, Greil R, Willborn KC, Wilhelm M, Debus J, Eble MJ, Sokler M, Ho A, Rank A, Ganser A, Trumper L, Bokemeyer C, Kirchner H, Schubert J, Kral Z, Fuchs M, Muller-Hermelink HK, Muller RP, Diehl V. Reduced treatment intensity in patients with early-stage Hodgkin's lymphoma. N Engl J Med. 2010 Aug 12;363(7):640-52. doi: 10.1056/NEJMoa1000067. PMID 20818855
- [Derived] Sasse S, Goergen H, Plutschow A, Boll B, Eichenauer DA, Fuchs M, Behringer K, Zijlstra JM, Greil R, Markova J, Topp MS, Meissner J, Neubauer A, Baues C, Engert A, Borchmann P, von Tresckow B. Outcome of Patients With Early-Stage Infradiaphragmatic Hodgkin Lymphoma: A Comprehensive Analysis From the German Hodgkin Study Group. J Clin Oncol. 2018 Sep 1;36(25):2603-2611. doi: 10.1200/JCO.2018.78.7192. Epub 2018 Jul 10. PMID 29989855
- [Derived] Boll B, Goergen H, Behringer K, Brockelmann PJ, Hitz F, Kerkhoff A, Greil R, von Tresckow B, Eichenauer DA, Burkle C, Borchmann S, Fuchs M, Diehl V, Engert A, Borchmann P. Bleomycin in older early-stage favorable Hodgkin lymphoma patients: analysis of the German Hodgkin Study Group (GHSG) HD10 and HD13 trials. Blood. 2016 May 5;127(18):2189-92. doi: 10.1182/blood-2015-11-681064. Epub 2016 Feb 1. PMID 26834240
- [Derived] Hay AE, Klimm B, Chen BE, Goergen H, Shepherd LE, Fuchs M, Gospodarowicz MK, Borchmann P, Connors JM, Markova J, Crump M, Lohri A, Winter JN, Dorken B, Pearcey RG, Diehl V, Horning SJ, Eich HT, Engert A, Meyer RM; Conducted by the NCIC Clinical Trials Group (Canada) and German Hodgkin Study Group (GHSG). An individual patient-data comparison of combined modality therapy and ABVD alone for patients with limited-stage Hodgkin lymphoma. Ann Oncol. 2013 Dec;24(12):3065-9. doi: 10.1093/annonc/mdt389. Epub 2013 Oct 11. PMID 24121121
- [Derived] Boll B, Gorgen H, Fuchs M, Pluetschow A, Eich HT, Bargetzi MJ, Weidmann E, Junghanss C, Greil R, Scherpe A, Schmalz O, Eichenauer DA, von Tresckow B, Rothe A, Diehl V, Engert A, Borchmann P. ABVD in older patients with early-stage Hodgkin lymphoma treated within the German Hodgkin Study Group HD10 and HD11 trials. J Clin Oncol. 2013 Apr 20;31(12):1522-9. doi: 10.1200/JCO.2012.45.4181. Epub 2013 Mar 18. PMID 23509310
- See also: Description of study in Gereman (Website of the Competence Network Malignant Lymphoma — http://www.lymphome.de/Gruppen/GHSG/